CLINICAL TRIAL: NCT01916109
Title: Phase II Study of Gemcitabine, Carboplatin, and Panitumumab (GCaP) as Neoadjuvant Chemotherapy in Patients With Muscle-Invasive Bladder Cancer
Brief Title: Study of Gemcitabine, Carboplatin, and Panitumumab (GCaP) as Neoadjuvant Chemotherapy in Patients With Muscle-Invasive Bladder Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-103
Record Dates: First submitted 2013-08-02; First posted 2013-08-05 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-01

CONDITIONS: Bladder Cancer
Keywords: Gemcitabine; Carboplatin; Panitumumab; (GCaP); radical cystectomy; 10-103
MeSH Terms: conditions — Urinary Bladder Neoplasms; Cone Dystrophy 3 | interventions — Gemcitabine; Carboplatin; Panitumumab; Cystectomy

ARMS (1):
- Gemcitabine, Carboplatin, and Panitumumab (GCaP) (Experimental): Patients will receive four cycles of GCaP administered every 21 days. Panitumumab will be administered intravenously at a dose of 9mg/kg on day 1. Gemcitabine 1,000 mg/m2 on day 1 and 8 and carboplatin AUC 4.5 on day 1 will be administered intravenously on a 21-day cycle. A total of four cycles of therapy will be administered at 21-day intervals followed by radical cystectomy.
  Interventions: Drug: Gemcitabine; Drug: Carboplatin; Drug: Panitumumab; Procedure: radical cystectomy

INTERVENTIONS:
Drug: Gemcitabine
Drug: Carboplatin
Drug: Panitumumab
Procedure: radical cystectomy

SUMMARY:
The purpose of this study is to find out if using the combination of standard chemotherapy (gemcitabine and carboplatin) plus this new drug (panitumumab) can help to shrink the tumor before the patient undergoes surgery for bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed muscle invasive transitional cell carcinoma of the bladder at MSKCC (Note: urothelial carcinoma invading into the prostatic stroma with no histologic muscle invasion is allowed, provided the extent of disease is confirmed via imaging and/or EUA.)
* Clinical stage T2-T4a N0/X M0 disease.
* Medically appropriate candidate for radical cystectomy as per MSKCC attending urologic oncologist
* Karnofsky Performance Status ≥ 80%
* Age ≥ 18 years of age
* Required Initial Laboratory Values:

Absolute neutrophil count ≥ 1500 cells/mm3

* Platelets ≥ 100,000 cells/mm3
* Hemoglobin ≥ 9.0g/dL
* Bilirubin ≤ 1.5 the upper limit of normal (ULN) for the institution
* Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN for the institution
* Alkaline phosphatase ≤ 2.5 x ULN for the institution
* Serum magnesium > 1.4 mEq/L
* Serum creatinine ≤ 2.0 mg/dL
* Cisplatin ineligibility based on one or more of the following criteria:

Estimated glomerular filtration rate (eGFR) 30-59 ml/min/1.73m2 using the CKD-EPI equation:(http://nephron.org/MDRD_GFR.cgi) :

eGFR = 141 x min(Scr/k, 1)a x max(Scr/k, 1)-1.209 x 0.993Age x 1.018 [if female] x 1.159 [if black] Scr is serum creatinine, k is 0.7 for females and 0.9 for males, a is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/k or 1, and max indicates the maximum of Scr/k or 1.

* Grade 2 sensory neuropathy
* Grade 2 hearing loss

  * Patients must provide a pretreatment saliva sample for genomic analysis.

Exclusion Criteria:

* Prior systemic chemotherapy (prior intravesical therapy is allowed)
* Serious intercurrent medical or psychiatric illness.
* Prior radiation therapy to the bladder.
* Concomitant use of any other investigational drugs
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, grade 2 or greater peripheral vascular disease, arterial thrombotic event, visceral arterial ischemia, cerebrovascular ischemia, transient ischemic attack, percutaneous transluminal angioplasty or stent, or unstable angina.

Symptomatic and/or serious uncontrolled arrhythmia

* Symptomatic congestive heart failure (NYHA class III or IVI)
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.
* History of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with the study participation or investigational product(s) administration or may interfere with the interpretation of the results.
* Major surgery requiring general anesthesia within 21 days or minor surgery within 14 days of study enrollment. Subjects must have recovered from surgery related toxicities.
* Pulmonary embolism, deep vein thrombosis, or other significant venous event ≤ 8 weeks before enrollment
* Known allergy or hypersensitivity to any component of the study treatment(s)
* Active infection requiring systemic treatment or any uncontrolled infections ≤14 days prior to enrollment.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
* Concurrent treatment on another clinical trial. Supportive care trials, surgical clinical trials or non-treatment trials, e.g. QOL, are allowed.
* Ongoing treatment with therapeutic doses of warfarin (low dose warfarin up to 2 mg po daily for thromboembolic prophylaxis is allowed).
* Pregnancy or breast-feeding. Patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy and for two (2) months following the last dose of panitumumab. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate. Male patients must be surgically sterile or agree to use effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-08; Primary Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean Bajorin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine, Carboplatin, and Panitumumab (GCaP): Gemcitabine, Carboplatin, and Panitumumab (GCaP) as Neoadjuvant Chemotherapy in Patients with Muscle-Invasive Bladder Cancer
Period: Overall Study
Arm/Group | Gemcitabine, Carboplatin, and Panitumumab (GCaP)
Started | 4
Completed | 3
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine, Carboplatin, and Panitumumab (GCaP)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate (<pT0)
Description: The absence of carcinoma (pT0 disease) and the absence of microscopic lymph node metastases (N0) on the final cystectomy specimen.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Gemcitabine, Carboplatin, and Panitumumab (GCaP)
Number analyzed (Participants) | 3
participants | 3

ADVERSE EVENTS:
Arm/Group | Gemcitabine, Carboplatin, and Panitumumab (GCaP)
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Carboplatin, and Panitumumab (GCaP) (N=4)
Wound dehiscence (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine, Carboplatin, and Panitumumab (GCaP) (N=4)
Anemia (Blood and lymphatic system disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Rash pustular (Skin and subcutaneous tissue disorders) | 1
Tremor (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes